CLINICAL TRIAL: NCT03502460
Title: Fluid Administration Limited by Lung Ultrasonography in the Operating Room: Correlation to Stroke Volume Variation (ORFALU)
Brief Title: Fluid Administration Limited by Lung Ultrasonography in the Operating Room: Correlation to Stroke Volume Variation.
Acronym: ORFALU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2017_843_0018
Record Dates: First submitted 2018-04-13; First posted 2018-04-18 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Surgery
Keywords: Lung ultrasonography; fluid administration; limitation; stroke volume variation; esophageal Doppler

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ORFALU (Other): Lung ultrasound consists of the application of a high-frequency ultrasound probe type Trans Thoracic Echography (ETT) on the anterior and lateral chest of the patient. Since air and bone do not pass through the US, it is the artefacts due to these structures that constitute ultrasound lung semiology.
  Esophageal Doppler is a means of monitoring cardiac output measuring stroke volume (SV).
  Interventions: Other: Operating Room Fluid Administration Lung Ultrasound

INTERVENTIONS:
Other: Operating Room Fluid Administration Lung Ultrasound — Use of lung ultrasound to limited fluid administration

SUMMARY:
The possibility of exploring the lungs by lung ultrasound, a non-invasive tool, is becoming increasingly popular for anesthesiologists. Recently, Lichtenstein has described the FALLS protocol (Fluid Administration Limited by Lung Sonography) which uses the potential of pulmonary ultrasound to evaluate early pulmonary overload due to fluid administration at a subclinical stage. Indeed, fluid administration can generate a sub-clinical interstitial syndrome that can be detected by passing from a profile A to a profile B in lung ultrasound. The transition from a profile A to a profile B therefore corresponds to the transition from a state of preload dependent to a state of preload independence. However, this tool has not been studied in the operating room. The main objective of this study will be to study the correlation between pulmonary ultrasound and SV variation measured by esophageal Doppler during fluid administration in patients with haemodynamic optimisation in the operating room during digestive, urological, gynecological and orthopedic surgeries. The main expected result is the following: good correlation between the absence of increased SV in the esophageal Doppler and the appearance of a B-profile lung ultrasound fluid administration in the operating room.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 ans
* inclusion criteria:
* Patient having a digestive, urological, gynecological, vascular or orthopedic surgery
* Haemodynamic optimisation requiring titration of the fluid administration
* Informed consent signed

Exclusion Criteria:

* Non-consent
* Chronic pulmonary pathology: COPD with pulmonary emphysema, pulmonary fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Apparition of Lines B at Lung Ultrasonography | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bar S, Yee C, Lichtenstein D, Sellier M, Leviel F, Abou Arab O, Marc J, Miclo M, Dupont H, Lorne E. Assessment of fluid unresponsiveness guided by lung ultrasound in abdominal surgery: a prospective cohort study. Sci Rep. 2022 Jan 25;12(1):1350. doi: 10.1038/s41598-022-05251-6. PMID 35079044